CLINICAL TRIAL: NCT04215848
Title: A Pilot Study of Efficacy of As-needed Budesonide/Formoterol Turbuhaler During Stepping Down Period From Step-3 in Adult Patients With Adequately Controlled Asthma
Brief Title: As-needed Budesonide/Formoterol Turbuhaler in Stepping Down Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Narongwit Nakwan, Head of Pulmonology, Hat Yai Medical Education Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 023/2562
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Asthma
Keywords: asthma; allergy
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- As-needed Budesonide/Formoterol (Experimental): As-needed Budesonide/Formoterol (160/4.5 ug)
  Interventions: Drug: Budesonide/Formoterol Fumarate 160 MCG-4.5 MCG Inhalation Powder
- Budesonide (Active Comparator): Budesonide (200 ug) twice daily
  Interventions: Drug: Budesonide 200Mcg Inhalation Powder

INTERVENTIONS:
Drug: Budesonide/Formoterol Fumarate 160 MCG-4.5 MCG Inhalation Powder — After the patients who have all criteria, they will be randomized to take Budesonide/formoterol (160/4.5 μg/d) as need when they have symptoms.
  Other Names: Symbicort Turbuhaler (160/4.5 ug)
  Arms: As-needed Budesonide/Formoterol
Drug: Budesonide 200Mcg Inhalation Powder — After the patients who have all criteria, they will be randomized to take Budesonide (200 μg) twice daily
  Other Names: Pulmicort Turbuhaler (200 ug)
  Arms: Budesonide

SUMMARY:
This study will evaluate the efficacy of as-needed Budesonide/formoterol Turbuhaler 160/4.5 µg/d in the period of step down in well controlled asthmatic patient comparing with standard maintenance therapy in step-2 management in asthma guildeline which is low dose inhaled corticosteroid.

DETAILED DESCRIPTION:
The study will measure the efficacy of as-needed low dose ICS/ LABA in well controlled asthmatic patient comparing with low dose ICS in step down circumstance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed as asthma at least 6 months.
2. Patients who have well controlled asthma by ACT > 23 and ACQ-7 < 0.75 at least 12 weeks with using budesonide/formoterol (160/4.5 μg/d) twice daily
3. Patient who not be taking oral bronchodilator such as montelukast, theophylline, doxophylline but accept for taking anti histamine and intranasal steroid.
4. Patients who able to do spirometry without contraindication.

Exclusion Criteria:

1. History of using systemic steroid previous 12 week and respiratory infection History of pulmonary tuberculosis with residual lung lesion by chest radiograph recent serious medical condition such as myocardial infarction, stroke, pneumonia etc.
2. History smoking less than 10 pack-years or be smoking
3. History of asthma exacabation previous 12 week

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Time to First moderate/severe asthma exacerbation rate or loss of asthma controlled | Patients will be followed for first moderate/severe asthma exacerbation rate or loss of asthma controlled (an estimated average duration of 24-48 weeks)
  Duration after the patients who has been randomised to developed asthma exacerbation or loss of asthma control that evaluation by Asthma Controlled Test (ACT)
Time to First moderate/severe asthma exacarbation rate | Patients will be followed for first moderate/severe asthma exacerbation rate (an estimated average duration of 24-48 weeks)
  Duration after randomisation until the patients will develop asthma exacerbation.
Time to First loss of asthma controlled | Patients will be followed for loss of asthma controlled (an estimated average duration of 24-48 weeks)
  Duration after randomisation until the patients will have a loss of asthma control evaluating by Asthma Controlled Test (ACT)
The ratio of asthma controlled to total number of participants | The ratio of asthma controlled to total number of participants at week 24th-48th.
  The ratio of participants who will be classified for asthma controlled to total number of participants by ACT score

SECONDARY OUTCOMES:
Change in lung function: FEV1%predicted | 24-48 weeks.
  Change from baseline in FEV1%predicted
Change in blood eosinophil count | 24-48 weeks.
  The change of absoluted eosinophil count after step down medication
Change in FENO | 48 weeks.
  The change of FENO after step down medication
Mean dose of inhaled steroid | 24-48 weeks.
  The amount of inhaled steroid dose throughout the study
Change in lung function: Peak expiratory flow | 24-48 weeks.
  Change from baseline in Peak expiratory flow

CONTACTS AND LOCATIONS:
Overall Officials: Narongwit Nakwan, M.D., Principal Investigator — HatYai Hospital
Locations (1):
- Hatyai Hospital, Hat Yai, Changwat Songkhla, Thailand